CLINICAL TRIAL: NCT05687123
Title: A Phase I Dose Escalation-Expansion Trial of Sunitinib Malate Plus Lutetium Lu 177 Dotatate (Lutathera) in Somatostatin Receptor Positive Pancreatic Neuroendocrine Tumors
Brief Title: Testing the Addition of Sunitinib Malate to Lutetium Lu 177 Dotatate (Lutathera) in Pancreatic Neuroendocrine Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-09321; NCI-2022-09321 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10479 (Other: Yale University Cancer Center LAO); 10479 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2023-01-14; First posted 2023-01-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Pancreatic Neuroendocrine Tumor; Pancreatic Neoplasm; Stage III Pancreatic Neuroendocrine Tumor AJCC v8; Stage IV Pancreatic Neuroendocrine Tumor AJCC v8; Unresectable Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Adenoma, Islet Cell; Pancreatic Neoplasms | interventions — Specimen Handling; lutetium Lu 177 dotatate; Magnetic Resonance Spectroscopy; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (sunitinib malate, lutetium Lu 177 dotatate) (Experimental): Patients receive sunitinib malate PO QD from day 1 of lutetium 177 dotatate therapy to 28 days after the last dose of lutetium 177 dotatate in the absence of unacceptable toxicity. Patients also receive lutetium Lu 177 dotatate IV over 30 minutes on day 1 of each cycle. Cycles repeat Q8W for 4 cycles in the absence of unacceptable toxicity. Patients undergo a CT scan and/or MRI throughout the trial. Patients also undergo a SSR PET/CT scan during screening and blood sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Lutetium Lu 177 Dotatate; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Sunitinib Malate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo a blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo a CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Lutetium Lu 177 Dotatate — Given IV
  Other Names: 177 Lu-DOTA-TATE; 177 Lu-DOTA-Tyr3-Octreotate; 177Lu-DOTA0-Tyr3-Octreotate; Lutathera; Lutetium (177Lu) Oxodotreotide; Lutetium Lu 177 DOTA(0)-Tyr(3)-Octreotate; Lutetium Lu 177-DOTA-Tyr3-Octreotate; lutetium Lu 177-DOTATATE; Lutetium Oxodotreotide Lu-177
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo a SSR PET/CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Sunitinib Malate — Given PO
  Other Names: SU 011248; SU 11248; SU-011248; SU-11248; SU011248; SU11248; sunitinib; Sutent

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of sunitinib malate in combination with lutetium Lu 177 dotatate in treating patients with pancreatic neuroendocrine tumors. Sunitinib malate is in a class of medications called kinase inhibitors and a form of targeted therapy that blocks the action of abnormal proteins called VEGFRs that signal tumor cells to multiply. This helps stop or slow the spread of tumor cells. Radioactive drugs, such as lutetium Lu 177 dotatate, may carry radiation directly to tumor cells and not harm normal cells. It is also a form of targeted therapy because it works by attaching itself to specific molecules (receptors) on the surface of tumor cells, known as somatostatin receptors, so that radiation can be delivered directly to the tumor cells and kill them. Giving sunitinib malate and lutetium Lu 177 dotatate in combination may be safer and more effective in treating pancreatic neuroendocrine tumors than giving either drug alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety and maximum tolerated dose (MTD) for the combination of sunitinib malate with lutetium Lu 177 dotatate in metastatic unresectable pancreatic neuroendocrine tumors (NETS).

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To assess objective response rate (ORR) of the combination by the Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.

III. To assess progression-free survival (PFS) and overall survival (OS) of the combination.

IV. To determine the duration of response (DOR) from the combination. V. To determine lutetium Lu 177 dotatate dosimetry in the combination. VI. To associate somatostatin receptor (SSR) positron emission tomography (PET) triage imaging with lutetium Lu 177 dotatate dosimetry.

VII. To assess the correlation of chromogranin A (CgA) with disease response in patients being treated with lutetium Lu 177 dotatate.

OUTLINE: This is a dose-escalation study of sunitinib malate followed by a dose-expansion study.

Patients receive sunitinib malate orally (PO) daily (QD) from day 1 of lutetium 177 dotatate therapy to 28 days after the last dose of lutetium 177 dotatate in the absence of unacceptable toxicity. Patients also receive lutetium Lu 177 dotatate intravenously (IV) over 30 minutes on day 1 of each cycle. Cycles repeat every 8 weeks (Q8W) for 4 cycles in the absence of unacceptable toxicity. Patients undergo a computed tomography (CT) scan and/or magnetic resonance imaging (MRI) throughout the trial. Patients also undergo a SSR PET/CT scan during screening and blood sample collection on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic, unresectable well- or moderately-differentiated pancreatic neuroendocrine tumors (PNETs) of any grade
* Patients with measurable disease appropriate for lutetium Lu 177 dotatate treatment as determined by positive screening with SSR PET/CT
* Patients may have disease progression on or intolerance of up to one line of systemic therapy other than somatostatin analog therapy. Prior and/or concurrent use of somatostatin analogs are allowed
* Patients who have documented disease progression per RECIST 1.1 within 12 months of initiation of the study protocol
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of sunitinib malate in combination with lutetium Lu 177 dotatate in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 1.5 institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 × institutional ULN
* Creatinine clearance > 50 ml/min OR Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2
* Hemoglobin > 8.0 g/dL
* White blood cell count > 2000/mL
* Serum calcium =< 12.0 mg/dL
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients must have blood pressure (BP) no greater than 140 mmHg (systolic) and 90 mmHg (diastolic) for eligibility. Initiation or adjustment of BP medication is permitted prior to study entry, provided that the average of three BP readings at a visit prior to enrollment is less than 140/90 mmHg
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression, as determined by a repeat imaging study at least 4 weeks following the completion of treatment. Patients with treated brain metastases must also be off steroids for at least 1 month and stable
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* The effects of lutetium Lu 177 dotatate and sunitinib malate on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because radionucleotides and anti-angiogenic agents are known to be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. All women of childbearing potential must have a negative pregnancy test prior to receiving sunitinib malate. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of lutetium Lu 177 dotatate and sunitinib malate administration

Exclusion Criteria:

* Patients who have not recovered from acute clinically significant adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib malate or lutetium Lu 177 dotatate
* Patients who require use of therapeutic doses of coumarin-derivative anticoagulants such as warfarin are excluded, although doses of up to 2 mg daily are permitted for prophylaxis of thrombosis. Note: Low molecular weight heparin is permitted provided the patient's prothrombin time (PT) international normalized ratio (INR) is =< 1.5
* Patients with any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain sunitinib tablets are excluded
* Patients with any of the following conditions are excluded:

  * Serious or non-healing wound, ulcer, or bone fracture
  * History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
  * Any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months prior to study entry
  * History of myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within 12 months prior to study entry
  * History of pulmonary embolism within the past 12 months
  * Class III or IV heart failure as defined by the New York Heart Association Class (NYHA) functional classification system
* Patients receiving any medications or substances that are strong CYP3A4 inhibitors within 7 days before dosing, or strong CYP3A4 inducers within 12 days before dosing, are ineligible as sunitinib is a major substrate of CYP3A4. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with a pre-existing thyroid abnormality who are unable to maintain thyroid function in the normal range with medication are ineligible
* Patients with uncontrolled intercurrent illness
* Pregnant women are excluded from this study because sunitinib malate is an anti-angiogenic agent and lutetium Lu 177 dotatate is a peptide receptor radionuclide therapy with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with sunitinib malate and lutetium Lu 177 dotatate, breastfeeding should be discontinued if the mother is treated with sunitinib malate and lutetium Lu 177 dotatate. Breastfeeding should be discontinued for 2.5 months following the last lutetium Lu 177 dotatate treatment. These potential risks may also apply to other agents used in this study
* Patients who have had prior treatment with sunitinib malate or lutetium Lu 177 dotatate therapy or other radiopharmaceuticals (including, but not limited to, metaiodobenzylguanidine [MIBG], yttrium-90 [Y-90], radioactive iodide [RAI]), as MIBG and RAI could potentially increase risk of myelodysplastic syndrome or irreversible hematologic toxicities
* Patients with left ventricular ejection fraction of 50% or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-12-14 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Within the first cycle (8 weeks)
  Dose-limiting toxicities (DLTs) during the first 8 weeks of the combination of sunitinib malate plus lutetium Lu 177 dotatate and incidence of treatment-emergent AEs during DLT observation period. DLTs will be defined as grade 3 or worse hematologic and non-hematologic toxicity that is considered clinically significant and at least possibly related to lutetium Lu 177 dotatate and sunitinib malate within the first cycle (8 weeks). Safety endpoints will be listed for each dose level and the tabulations of adverse events will also be produced by severity and by relationship to study drug

SECONDARY OUTCOMES:
Objective response (ORR) | Up to 4 weeks
  ORR defined as the percentage of patients who achieve complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. For efficacy data in the expansion cohort, ORR and its 95% confidence interval will be calculated.
Duration of response | The time from first documentation of response (CR or PR) until the time of first documentation of disease progression by RECIST v1.1, assessed up to 4 weeks
  The change over-time as well as the difference between sub-groups (i.e., toxicity by Common Terminology Criteria for Adverse Events [CTCAE], tumor response by RECIST 1.1, etc.) will be summarized using descriptive statistics and presented graphically.
Progression-free survival (PFS) | The time from first dose to the earlier date of assessment of progression or death by any cause, assessed up to 4 weeks
  The distribution of PFS will be described using Kaplan-Meier product limit methods. The change over-time as well as the difference between sub-groups (i.e., toxicity by CTCAE, tumor response by RECIST 1.1, etc.) will be summarized using descriptive statistics and presented graphically.
Overall survival (OS) | From the date of first dose to the date of death by any cause, assessed up to 4 weeks
  The distribution of OS will be described using Kaplan-Meier product limit methods. The change over-time as well as the difference between sub-groups (i.e., toxicity by CTCAE, tumor response by RECIST 1.1, etc.) will be summarized using descriptive statistics and presented graphically.
Intensity of tumor uptake | Up to 4 weeks
  Intensity of tumor uptake on pre-treatment somatostatin receptor (SSR) positron emission tomography (PET) and post-lutetium Lu 177, as well as the dosimetry imaging. The organ dosimetry will be summarized using descriptive statistics at each time point. The correlation between intensity of tumor uptake on pre-treatment SSR PET and post-lutetium Lu 177, as well as the dosimetry imaging will also be described using Spearman or Pearson correlation coefficient.
Chromogranin A levels | Up to 4 weeks
  Chromogranin A levels will be measured and chromogranin A responses will be defined as 50% or greater reduction from baseline or normalization per RADIANT-1 study. Chromogranin A levels and responses will be summarized using descriptive statistics. Responses will be correlated with radiographic responses using contingency tables.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Trikalinos, Principal Investigator — Yale University Cancer Center LAO
Locations (10):
- United States (9):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Memorial Hospital East, Shiloh, Illinois
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
"NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page."
URL: https://grants.nih.gov/policy/sharing.htm